CLINICAL TRIAL: NCT01436188
Title: A Biomarker Study to Measure CSF Proteins Upon Application of an Indwelling Lumbar Catheter for 36 Hours in Elderly Healthy Subjects and Subjects With Mild Cognitive Impairment or Alzheimer's Disease
Brief Title: A Study to Measure CSF Proteins in Elderly Healthy Volunteers and Volunteers With Mild Cognitive Impairment or Alzheimer's Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CR100658; NOCOMPOUNDEDI0001 (Other: Janssen Research & Development, LLC); 2011-003525-94 (EudraCT Number)
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Healthy; Alzheimer Disease
Keywords: Biological Markers; Healthy Volunteer; Alzheimer's Disease (AD); Mild Cognitive Impairment (MCI); Cerebrospinal fluid (CSF); CSF proteins
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Ibuprofen

ARMS (5):
- 001 (Healthy Elderly Cohort 1) (Other): standard frequent CSF sampling procedure for 36 hours
  Interventions: Procedure: Standard CSR sampling procedure
- 002 (Healthy Elderly Cohort 2) (Other): an alternative frequency of CSF sampling procedure for 36 hours
  Interventions: Procedure: Alternate frequency CSR sampling procedure
- 003 (Healthy Elderly Cohort 3) (Other): standard frequent CSF sampling procedure on Day 1 for 36 hours with 800 mg Ibuprofen administered on Day 1
  Interventions: Procedure: Standard frequent CSR sampling procedure with 800 mg ibuprofen
- 004 (Elderly Volunteers with MCI or AD) (Other): standard CSF sampling procedure for 36 hours
  Interventions: Procedure: Standard CSR sampling procedure
- 005 (Healthy Eldely Cohort 5) (Other): an alternative lower frequency of CSF sampling in comparison to Cohort 1
  Interventions: Procedure: Alternative lower frequency CSR sampling procedure

INTERVENTIONS:
Procedure: Standard CSR sampling procedure — standard frequent CSF sampling procedure for 36 hours
  Arms: 001 (Healthy Elderly Cohort 1)
Procedure: Alternate frequency CSR sampling procedure — an alternative frequency of CSF sampling procedure for 36 hours
  Arms: 002 (Healthy Elderly Cohort 2)
Procedure: Standard frequent CSR sampling procedure with 800 mg ibuprofen — standard frequent CSF sampling procedure on Day 1 for 36 hours with 800 mg Ibuprofen administered on Day 1
  Arms: 003 (Healthy Elderly Cohort 3)
Procedure: Standard CSR sampling procedure — standard frequent CSF sampling procedure for 36 hours.
  Arms: 004 (Elderly Volunteers with MCI or AD)
Procedure: Alternative lower frequency CSR sampling procedure — an alternative lower frequency of CSF sampling procedure in comparison to Cohort 1 for 36 hours
  Arms: 005 (Healthy Eldely Cohort 5)

SUMMARY:
The purpose of this study is to investigate changes of cerebral spinal fluid (CSF) proteins over time using continuous CSF sampling for 36 hours in elderly healthy volunteers and volunteers with mild cognitive impairment or Alzheimer's Disease.

DETAILED DESCRIPTION:
This is a study to measure specific proteins in the cerebral spinal fluid (CSF) of healthy elderly volunteers and volunteers with mild cognitive impairment (MCI) or Alzheimer's Disease (AD). No investigational medical drug will be given to volunteers during their participation in this study. Healthy elderly volunteers will be enrolled in Part A of the study and will be randomized (assigned by chance) to 1 of 4 cohorts (groups); each cohort of volunteers will undergo a different type of CSF sampling procedure (a standard frequent CSF sampling procedure, an alternative frequency of CSF sampling procedure, or the standard frequent CSF sampling procedure with 800 mg ibuprofen administered to volunteers on Day 1, or an alternative lower frequency of CSF sampling in comparison to Cohort 1) and will have blood samples collected. Volunteers with MCI or AD will be enrolled in Part B of the study and will undergo 1 CSF sampling procedure (ie, the standard frequent CSF sampling procedure). In addition, all volunteers enrolled who consent (agree) to the pharmacogenomic component of the study, will have a blood sample collected that will allow for genetic research to help understand the link between Alzheimer's Disease biomarker profiles and specific genotypes and to have their DNA samples stored for future genetic research related to CSF proteins and Alzheimer's Disease. Participation in the pharmacogenomic research is optional for volunteers enrolled in Part A Cohort 1 to 3 but required for volunteers enrolled in Part A Cohort 5 and Part B. Participation in the DNA storage component is optional and refusal to participate will not result in ineligibility for the main part of the study. There will be no blinding in this study (ie, volunteers will know the CSF sampling procedure being performed on them). CSF and blood samples will be collected over a period of 36 hours and the maximum duration of the study will be no more than 6 weeks. During the study, volunteers will be monitored to evaluate the safety and tolerability of the CSF sampling procedures.

ELIGIBILITY:
Inclusion Criteria:

* Healthy elderly Volunteers (Part A: age range 55 to 85 years of age, inclusive) and Volunteers with AD or MCI and a typical AD biomarker signature (Part B: age range 50 to 90 years of age, inclusive), with a body mass index (BMI) between 18 and 35 kg/m2 (inclusive) who satisfy the additional inclusion criteria specified in the study protocol will be eligible for enrollment in this study

Exclusion Criteria:

* Has a clinically significant abnormal physical or neurological examination (including fundoscopy), vital signs or 12-lead electrocardiogram (ECG) at screening
* Has a relevant history of lower back pain or scoliosis and/or major (lumbar) back surgery (microdiscectomy is allowed)
* Has a history of spontaneous, prolonged or severe bleeding with unclear origin
* Has a history of epilepsy or fits or unexplained black-out
* has any other exclusion criteria as specified in the study protocol

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-09; Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Measurement of CSF proteins | 36 hours
  The changes in CSF proteins over 36 hours after lumbar introduction of a spinal catheter will be investigated.

SECONDARY OUTCOMES:
The number of volunteers with adverse events | Up to 6 weeks
  The number and type of adverse events reported will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (3):
- Antwerp, Belgium
- Netherlands (2):
  - Groningen
  - Leiden

REFERENCES:
- [Derived] Van Broeck B, Timmers M, Ramael S, Bogert J, Shaw LM, Mercken M, Slemmon J, Van Nueten L, Engelborghs S, Streffer JR. Impact of frequent cerebrospinal fluid sampling on Abeta levels: systematic approach to elucidate influencing factors. Alzheimers Res Ther. 2016 May 19;8(1):21. doi: 10.1186/s13195-016-0184-z. PMID 27206648